CLINICAL TRIAL: NCT02190578
Title: Clinical Performance of Reveal G4 Rapid HIV-1 Antibody Test for the Detection of HIV-1 Antibodies in Fingerstick and Venous Whole Blood Samples
Brief Title: Clinical Performance of Reveal G4 Rapid HIV-1 Antibody Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MedMira Laboratories Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MCP005
Record Dates: First submitted 2014-07-11; First posted 2014-07-15 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2014-07

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Diagnostic: Reveal G4 (Experimental): Subjects tested with investigational devices and approved comparator assay algorithms for HIV
  Interventions: Device: Reveal G4

INTERVENTIONS:
Device: Reveal G4 — All subjects tested with the investigational device, Reveal G4, plus with an algorithm of approved assays for HIV.
  Other Names: Reveal Rapid HIV-1 Antibody Test

SUMMARY:
To determine the efficacy of an improved rapid diagnostic test using venous whole blood and fingerstick whole blood. The clinical performance of Reveal G4 Rapid HIV-1 Antibody Test will be determined by comparing the results with patient infected status for HIV-1 (human immunodeficiency virus type 1).

The study will consist of a single one-hour visit, at which time blood samples will be collected and tested with the investigational device (Reveal G4) and FDA approved comparator assays for detection of HIV-1 antibodies.

DETAILED DESCRIPTION:
This clinical trial is a multi-center study to assess the performance characteristics of a rapid in vitro diagnostic assay, the Reveal G4 Rapid HIV-1 Antibody Test (Reveal G4). Specifically, the objective of this study is to determine the sensitivity and specificity of Reveal G4 in finger stick and venous whole blood, relative to FDA approved reference assays for the detection of HIV-1 antibodies.

Approximately 1500-2000 subjects in total will be enrolled in the study across all sites, into three different study populations. Population 1 will be comprised of at least 500 subjects from a population at risk of infection with HIV. Population 2 will be comprised of at least 500 subjects that are known HIV positive individuals. Population 3 will be comprised of at least 500 subjects from a population at low risk of HIV infection. Reveal G4 will be used to test fingerstick whole blood and venous whole blood samples from all study subjects. For enrolled subjects in Populations 1 and 3, who are of unknown HIV antibody status, a plasma sample prepared from the venous whole blood sample will also be tested with an algorithm of FDA-approved assays for the detection of HIV-1 antibodies. For Population 2 subjects who are known HIV-positive individuals, results of previous HIV tests will be obtained from the subjects' medical records. The sensitivity and specificity of Reveal G4 will be determined in fingerstick and venous whole blood relative to HIV-1 antibody status as determined by an algorithm of FDA-approved assays.

The primary analysis will involve comparison of Reveal G4 results for anti-HIV-1 in each sample matrix (fingerstick whole blood and venous whole blood) with the subject's HIV-1 antibody status as determined by FDA-approved assays. Based on the above, the sensitivity and specificity of Reveal G4 will be determined with corresponding two-sided 95% confidence intervals for both fingerstick and venous whole blood.

ELIGIBILITY:
Inclusion Criteria:

* All subjects must be at least 18 years of age, able to sign consent form, complete the risk assessment questionnaire, and provide the required blood samples: fingerstick sample (1 drop), venous whole blood sample (1 K2 EDTA tube).

  * Population 1 - Individuals at risk of HIV infection (n ≥ 500) Subjects must meet have at least one risk factor for infection with HIV
  * Population 2 - Known HIV-1 positive individuals (n ≥ 500) Subjects must be a known HIV-positive individual (previous positive HIV test result)
  * Population 3 - Individuals at low risk of HIV infection (n ≥ 500) Subjects must not have any risk factors for infection with HIV

Exclusion Criteria:

* Subjects do not meet inclusion criteria

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1649 (Actual)
Dates: Start 2014-07; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Determine clinical performance of Reveal G4 | At single study visit (one hour)
  To determine the clinical performance of Reveal G4 with fingerstick and venous whole blood relative to the HIV-1 infected status of the patient

CONTACTS AND LOCATIONS:
Overall Officials: Fabienne Laraque, MD, Principal Investigator — New York City Department of Health and Mental Hygiene; Peter Kerndt, MD, Principal Investigator — University of Southern California - Los Angeles; Cheryl Berne, MD, Principal Investigator — Biological Specialties Corporation; Anthony LaMarca, MD, Principal Investigator — Therafirst Medical Center
Locations (4):
- United States (4):
  - Preventive Medicine, University of Southern California (Los Angeles), Los Angeles, California
  - Therafirst Medical Center, Fort Lauderdale, Florida
  - New York City Department of Health and Mental Hygiene, Queens, New York
  - Biological Specialty Corporation, Reading, Pennsylvania